CLINICAL TRIAL: NCT02669732
Title: A Phase 2, Randomized, Placebo-controlled, Double-blind, Crossover Study of DS-8500a to Evaluate the Effects on Pancreatic Beta Cell Function in Japanese Patients With Type 2 Diabetes Mellitus.
Brief Title: An Exploratory Study of DS-8500a on Beta Cell Function Using Hyperglycemic Clamp
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Daiichi Sankyo Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Daiichi Sankyo (Industry)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DS8500-A-J205
Record Dates: First submitted 2016-01-27; First posted 2016-02-01 (Estimated); Last update posted 2019-02-12 (Actual); Status verified 2016-12

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Type 2 Diabetes Mellitus; Adult; Developmental Phase II
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — firuglipel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- DS-8500a 75 mg once daily (QD) (Experimental): tablets, orally, once daily for up to 28 days
  Interventions: Drug: DS-8500a
- Placebo (Placebo Comparator): tablets, orally, once daily for up to 28 days
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: DS-8500a — tablets
  Arms: DS-8500a 75 mg once daily (QD)
Drug: placebo — tablets
  Arms: Placebo

SUMMARY:
The objective of the study is to evaluate change in insulin secretory capacity in patients with type 2 diabetes mellitus as determined by hyperglycemic clamp after a 28-day oral administration of DS-8500a at 75 mg in a placebo-controlled, 2 × 2 crossover study. In addition, safety of this regimen will be examined in this study.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥ 20 years at the time of informed consent
* Japanese patients with type 2 diabetes
* Patients who have HbA1c ≥ 7.0% and < 9.0%

Exclusion Criteria:

* Patients with type 1 diabetes mellitus or with a history of diabetic coma, precoma, or ketoacidosis
* Patients receiving or requiring treatment with insulin
* Patients with a body mass index (BMI) of < 18.5 kg/m2 or ≥ 35.0 kg/m2
* Patients with clinically evident renal impairment (estimated glomerular filtration rate [eGFR] of < 45 mL/min per 1.73 m2) or clinically significant renal disease
* Patients with fasting plasma glucose ≥ 240 mg/dL

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2016-01; Primary Completion 2016-08 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
First-phase and Second-phase secretion Insulin | Baseline to Day 28 (Period 1 and 2)
  First-phase and Second-phase secretion Insulin Baseline to Day 28 (Period 1 and 2)
First-phase and Second-phase secretion C-peptide | Baseline to Day 28 (Period 1 and 2)
  First-phase and Second-phase secretion (C-peptide)

SECONDARY OUTCOMES:
M value | Baseline to Day 28 (Period 1 and 2)
  M value：Mean of Glucose Infusion Rate from 90 to 120 min
M/I value | Baseline to Day 28 (Period 1 and 2)
  M/I value：M value / steady-state Insulin
Disposition Index | Baseline to Day 28 (Period 1 and 2)
  Disposition Index：Product of M value and First-phase secretion
Number and severity of Adverse Events | Day 28 (Period 1 and 2)
plasma concentration of DS-8500a | Day 28 (Period 1 and 2)

CONTACTS AND LOCATIONS:
Overall Officials: Hirotaka Watada, MD, PhD, Principal Investigator — Juntendo University
Locations (1):
- SOUSEIKAI Hakata Clinic, Hakata-ku, Fukuoka, Japan

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/